CLINICAL TRIAL: NCT00981552
Title: Dosimetric Planning Study Comparing IMRT and 4-field Radiotherapy for Definitive Treatment of Cancer of the Cervix
Brief Title: Dosimetric Planning Study Comparing Intensity Modulated Radiotherapy (IMRT) and 4-field Radiotherapy for Definitive Treatment of Cancer of the Cervix
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr Gillian Thomas, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMRTCC
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Cervix Cancer
Keywords: Cervix Cancer; IMRT; Organ Motion; Target Definition
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cervix Cancer (Other): Patients treated with cervical cancer in 2008 at Sunnybrook Odette Cancer Centre
  Interventions: Radiation: IMRT planning; Radiation: 4-Field Radiation Planning

INTERVENTIONS:
Radiation: IMRT planning
Radiation: 4-Field Radiation Planning

SUMMARY:
A theoretical planning study to compare the normal tissue irradiation when using intensity modulated radiotherapy (IMRT) as opposed to standard radiotherapy for the definitive treatment of cervical cancer.

DETAILED DESCRIPTION:
Radiotherapy in combination with chemotherapy is the standard treatment of locally advanced cervix cancer, however with traditional techniques large volumes of bowel and bladder are irradiated causing short-term and long-term genito-urinary and gastro-intestinal side effects. IMRT has the potential to conform precisely to the target and spare normal tissues and reduce side effects. However because there are large dose gradients there is the potential to miss the target due to organ motion. Recent studies have documented organ motion and will be used to define the target. Approximately 60 planning scans, previously used to treat patients with cervix cancer, will be used to replan using an IMRT technique and differences in doses to tumour and normal tissues compared.

ELIGIBILITY:
Inclusion Criteria:

* last 60 patients treated definitively for cervical cancer at Sunnybrook Odette Cancer Centre

Exclusion Criteria:

* no imaging and no anatomical description of disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Reduction in dose to organs at risk | 6 months

SECONDARY OUTCOMES:
Target Coverage | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Thomas, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada